CLINICAL TRIAL: NCT01407770
Title: Impact of Genomics and Exposures on Disparities in Breast Cancer Radiosensitivity
Brief Title: Genetic Susceptibility to Radiation-Induced Skin Reactions in Racial/Ethnic Groups of Patients With Breast Cancer
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: IRB00011809; U10CA081851 (NIH); REBACCCWFU97609 (Other: NCI)
Record Dates: First submitted 2011-07-30; First posted 2011-08-02 (Estimated); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Breast Cancer; Cognitive Ability, General; Fatigue; Pain; Psychosocial Deprivation; Radiation Toxicity; Skin Abnormalities
Keywords: radiation toxicity; skin reactions secondary to radiation therapy; pain; fatigue; psychosocial effects of cancer and its treatment; depression; cognitive/functional effects; stage IA breast cancer; stage IB breast cancer; stage II breast cancer; stage IIIA breast cancer; ductal breast carcinoma in situ
MeSH Terms: conditions — Breast Neoplasms; Fatigue; Pain; Radiation Injuries; Skin Abnormalities; Depression; Carcinoma, Intraductal, Noninfiltrating | interventions — Gene Expression Profiling; Enzyme-Linked Immunosorbent Assay; Flow Cytometry; Chemotherapy, Adjuvant; Radiotherapy, Conformal; Radiotherapy, Intensity-Modulated

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — blood and urine samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Genetic: DNA analysis — Genetic
Genetic: gene expression analysis — Genetic
Other: enzyme-linked immunosorbent assay — Genetic
Other: flow cytometry — Genetic
Other: laboratory biomarker analysis — Genetic
Other: questionnaire administration — Genetic
Procedure: adjuvant therapy — Genetic
Procedure: assessment of therapy complications — Genetic
Procedure: quality-of-life assessment — Genetic
Radiation: 3-dimensional conformal radiation therapy — Genetic
Radiation: breast irradiation — Genetic
Radiation: external beam radiation therapy — Genetic
Radiation: hypofractionated radiation therapy — Genetic
Radiation: intensity-modulated radiation therapy — Genetic
Radiation: whole breast irradiation — Genetic

SUMMARY:
RATIONALE: Radiation therapy uses high-energy x rays to kill tumor cells. Radiation therapy may cause skin reactions when patients are exposed to high-energy x rays. Studying the genetic pattern of patients before and after radiation therapy may help doctors prevent toxicity and plan the best treatment.

PURPOSE: This clinical trial studies genetic susceptibility to radiation-induced skin reactions in racial/ethnic groups of patients with breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* To develop and validate prediction biomarkers for radiation therapy (RT)-induced acute and chronic skin reactions and quality of life in five racial/ethnic groups of breast cancer patients, Whites*, Black/African Americans, Hispanic/Latinos, Asians/Native Hawaiians/Pacific Islanders, and American Indians/Alaskan Natives. NOTE: *This stratum is closed as of April 25, 2012.
* To develop polygenic models of RT-induced skin reactions with a comprehensive evaluation of genome-wide nonsynonymous single nucleotide polymorphisms (nsSNPs).
* To evaluate the levels of DNA damage (Comet assay) and radiosensitivity (Cell Cycle G2 Delay assay) in lymphocytes before and after RT.
* To test the effect of gene-gene and gene-smoking interactions on RT-induced skin reactions.
* To assess race-ethnic differences in RT-induced skin reactions, DNA damage, and radiosensitivity and to determine if the gene effects are consistent across race-ethnicity (gene-race/ethnic interactions).

OUTLINE: This is a multicenter study. Patients are stratified according to race/ethnicity (Whites* vs Black/African Americans vs Hispanic/Latinos vs Asians/Native Hawaiians/Pacific Islanders vs American Indians/Alaskan Natives). NOTE: *This stratum is closed as of April 25, 2012.

Patients undergo adjuvant radiotherapy after breast-conserving surgery.

Blood and urine samples are collected at baseline and last day of radiotherapy for genotyping, DNA damage, cell cycle assays, urine cotinine, inflammatory immune response biomarkers, and tumor-killing activity by BeadArray System, Comet assay, flow cytometry-based assay, Cell-Cycle G2 Delay Assay, Oxygen Radical Absorbance Capacity (ORAC) assay, and ELISA.

Patients are assessed for acute toxicity by research staff using the ONS Criteria for Radiation-Induced Acute Skin Toxicity at baseline, week 3, and at 1 and 2 months after radiotherapy. Patients are also assessed for chronic toxicity by research staff using the Chronic skin toxicity questionnaire (RTOG SOMA Criteria for RT- Induced Breast/Chest Wall Late Skin Toxicity) at 6 and 12 months after completion of radiotherapy. Photographs of the breast, chest wall, and contralateral breast are also taken at baseline, week 3, last day of radiotherapy, and at 1, 2, 6, and 12 months after completion of radiotherapy.

Patients complete the Breast Cancer Risk Study Questionnaire, the Functional Assessment of Cancer Therapy Breast (FACT-B), the Modified Skindex, and the B39 Quality-of-Life (QOL) Questionnaire at baseline, last day of radiotherapy, and at 1, 2, 6, and 12 months after radiotherapy.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Female patients newly diagnosed with breast carcinoma including ductal carcinoma in situ (DCIS)

  * Stage 0-IIIA disease
* Status post-lumpectomy, -quadrantectomy, or -mastectomy
* Plan to receive adjuvant radiation to the whole breast or chest wall and/or regional lymph nodes
* No sites that cannot send blood/urine specimens to Wake Forest by overnight (next day) express shipping

PATIENT CHARACTERISTICS:

* *This stratum is closed as of April 25, 2012.
* No patients who do not understand English and are unable to complete form with assistance

PRIOR CONCURRENT THERAPY:

* Total dose > 40 Gy, dose per fraction > 1.8 - 2.0 Gy, use of 2D, 3D-conformal, or intensity-modulated radiation therapy (IMRT) treatment techniques allowed; a daily fraction of 2.7 Gy to the whole breast is suggested for hypofractionated regimens
* Concurrent and sequential boost techniques are allowed for both standard and hypofractionated regimens
* Adjuvant hormonal therapy will be allowed prior to, during, and/or after radiotherapy (RT) at the discretion of a medical oncologist
* Targeted therapies, such as Herceptin, will be allowed prior to, during, and/or after RT at the discretion of the medical oncologist
* No prior radiation to the involved breast or chest wall
* No concurrent chemotherapy
* No patients who underwent breast reconstruction following mastectomy

  * Placement of tissue expanders and implants are not allowed
* No patients who have undergone MammoSite® or any other form of brachytherapy as well as those who will be treated with skin-sparing IMRT
* Patients may not be concurrently enrolled in a protocol that involves treatment of the skin, i.e., applying lotions/moisturizers

  * Protocols that do not involve treatment of the skin are allowed

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Race/ethnicity to include Whites*, Black/African Americans (AA), Hispanic/Latinos, Asians/Native Hawaiians/Pacific Islanders, and Native American or Alaskan
Sampling Method: Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2011-09-20 (Actual); Primary Completion 2014-08-26 (Actual); Study Completion 2014-08-26 (Actual)

PRIMARY OUTCOMES:
Occurrence of RT-induced early adverse skin reaction (EASR) | 2 months
  The primary endpoint is RT-related skin reactions which for consistency and clarity across the study we will use the term "Early Adverse Skin Reaction" (EASR). Skin reactions will be assessed at 4 time points from the start of radiotherapy through 2 months of the post radiotherapy follow-up period. The Modified ONS Criteria for Radiation-Induced Acute Skin Toxicity will be used for classification of EASRs related to the skin. The primary outcome variable will be the occurrence (or not) of RT-induced EASR defined as a grade 4 or higher toxicity (based on the ONS criteria) during the 2 months of the follow-up period of the study.

SECONDARY OUTCOMES:
Quality of life as measured by FACT-B | 12 months
  Quality of life will be assessed using the FACT-B, a modification of the Skindex-16, and a modified version of the NSABP B39 Quality of Life metric.

CONTACTS AND LOCATIONS:
Overall Officials: James J. Urbanic, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Comprehensive Cancer Center, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Hu JJ, Urbanic JJ, Case LD, Takita C, Wright JL, Brown DR, Langefeld CD, Lively MO, Mitchell SE, Thakrar A, Bryant D, Baglan K, Strasser J, Baez-Diaz L, Lesser GJ, Shaw EG. Association Between Inflammatory Biomarker C-Reactive Protein and Radiotherapy-Induced Early Adverse Skin Reactions in a Multiracial/Ethnic Breast Cancer Population. J Clin Oncol. 2018 Aug 20;36(24):2473-2482. doi: 10.1200/JCO.2017.77.1790. Epub 2018 Jul 10. PMID 29989859